CLINICAL TRIAL: NCT00990418
Title: Bioequivalence Between Integrated E-TRANS (Fentanyl) System and Separated (Two-Part) E-TRANS (Fentanyl) System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Senior Director, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR013654
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; E-TRANS System, fentanyl HCl System; E-TRANSS (fentanyl HCl) System; Acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Divorce; Drug Delivery Systems

INTERVENTIONS:
Drug: Separated (Two Part) E-TRANS (fentanyl HCl) System; Integrated E-TRANS (fentanyl HCl) System

SUMMARY:
The purpose of this study is to confirm that the two forms of the device the Integrated E-TRANS (fentanyl HCl) system and the Separated (Two-Part) E-TRANS (fentanyl HCl) System provide the equivalent blood levels of medication (fentanyl HCL).

DETAILED DESCRIPTION:
The objective of this study is to establish bioequivalence between the Integrated E-TRANS (fentanyl HCl) System and the Separated (Two-Part) E-TRANS (fentanyl HCl) System. The target indication is the short-term management of acute postoperative pain in adult patients requiring opioid analgesia during hospitalization. This is a single-center, open-label (all people involved know the identity of the intervention), randomized, 2-period, 2-treatment, 2-sequence, crossover (participants will receive different interventions sequentially during the study) interventions study. Each volunteer will be randomly assigned to a sequence. There will be a washout period of 6 to 14 days between treatments. Volunteers will remain at the study site during fentanyl treatments and for the 34 hours following completion of each treatment. Approximately 60 healthy volunteers will be enrolled to ensure that 40 volunteers have completed pharmacokinetic evaluations in both treatments. Each volunteer will receive both Treatment A and Treatment B (either Treatment A followed by Treatment B or Treatment B followed by Treatment A.) Treatment A is 80 consecutive doses of Ontegrated E-TRANS (fentanylHCL) 40mcg System, each delivered over 10 minutes for a total delivery time of over 13.33 hours. Treatment B is 80 consecutive doses of Separated (Two-Part) E-TRANS (fentanyl HCL) 40 mcg System, each delivered over 10 minutes, for a total deliver time of over 13.33 hours. Blood samples for pharmacokinetic analysis (analysis of the amount of drug in the blood at specific time points) will be collected from each volunteer during all fentanyl treatments and up to 34 hours after termination of each treatment. The skin site to which an E-TRANS (fentanyl HCl) System has been applied will be monitored for the development of topical (skin irritation) adverse events at 1 and 24 hours after removal of the system(s). Safety evaluations to be performed include adverse event monitoring, laboratory assessments, alcohol testing, serum pregnancy testing for women of child-bearing potential, urine drug screening, physical examination, electrocardiogram, continuous pulse oximetry to monitor oxygen saturation, respiratory rate, blood pressure, heart rate, respiratory rate, and temperature. The study will continue for up to approximately 3 weeks, including the washout periods of 6 to 14 days in between treatments, excluding the screening period. Treatment A: Integrated E-TRANS (fentanyl HCl) 40 mcg System 80 consecutive doses, each delivered over 10 minutes over 13.33 hours Treatment B: Separated (Two-Part) E-TRANS (fentanyl HCl) 40 mcg System 80 consecutive doses, each delivered over 10 minutes over 13.33 hours. Volunteers will be randomly assigned to either receive either Treatment A followed by Treatment B or Treatment B followed by Treatment A.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (of 18.0 to 28.0 kg/m2 at screening
* Healthy based on medical history, physical examination, blood chemistry, blood count, urinalysis, and electrocardiogram
* Blood pressure between 90 to 139 mmHg systolic (inclusive) and 50 to 89 mmHg diastolic (inclusive) after sitting for 5 minutes

Exclusion Criteria:

* Evidence of clinically significant hepatic, reproductive, gastrointestinal, renal, hematologic, pulmonary, neurologic, respiratory, endocrine, or cardiovascular system abnormalities, psychiatric disorders or acute infection
* Patients with confirmed screening QTc interval >450 msec or a history of additional risk factors for torsades de pointes, or the use of other medications that are currently being taken that prolong the QT/QTc interval (measure of electric conduction in the heart by ECG test)
* Patients who have supine-to-standing blood pressure decrease of >20 mmHg systolic or >10 mmHg diastolic after standing for 3 minutes or have symptoms of lightheadedness, dizziness, or fainting upon standing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the bioequivalence of the Separated (Two-Part) E-TRANS (fentanyl HCl) System and the Integrated E-TRANS (fentanyl HCl) System | 0 (predose), 0.5, 1.0, 2.0, 4.0, 6.0, 8.0, 10.0, 11.0, 12.5, 13.33, 13.5, 14.0, 15.0, 16.0, 18.0, 20.0, 24.0, 27.0, 30.0, 36.0, and 47.0 hours after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA